CLINICAL TRIAL: NCT02525978
Title: Relationship Between Heart Rate Variability and Emotional Experience in Healthy and Depressed Adults
Brief Title: Heart Rate Variability in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Andrea Crowell, Senior Associate, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00082047
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Major Depressive Disorder
Keywords: Heart Rate
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Controls (Experimental): Healthy controls will complete the video task and imaginal task in one session
  Interventions: Behavioral: Video Task; Other: Imaginal Task
- Depressed + Ketamine (Experimental): Subjects with major depressive disorder (MDD) who are scheduled to receive ketamine infusions will complete the video task and imaginal task twice. The first visit will be before any ketamine treatment. The second visit will be within 1 week after first ketamine infusion. This is NOT at treatment study. Study inclusion is open to participants with MDD who are already planning to receive ketamine treatment at Emory. No treatment is offered through this study.
  Interventions: Behavioral: Video Task; Other: Imaginal Task

INTERVENTIONS:
Behavioral: Video Task — Subjects are asked to watch a series of six two-minute video clips. The video clips are designed to induce sad or happy emotions or no emotion (neutral) and are taken from movies, documentaries, or instructional videos. There are two videos for each emotion condition. Videos and fixation cross screens are viewed on a laptop computer. In between video clips, patients are asked to quietly look at a fixation cross for one minute, describe their emotional reaction to the video for up to one minute, then again attend to a fixation cross for one minute. A video recording of the frontal view of the participant's face will be made during task performance.
Other: Imaginal Task — Subjects are asked to think about happy or sad memories for 2 minutes. Subjects are asked to imagine performing neutral tasks, such as buying groceries. Subjects are then asked to think about a memory that makes them feel angry. A video recording of the frontal view of the participant's face will be made during task performance.

SUMMARY:
The purpose of this study is to understand if there is a relationship between the way that emotions are regulated by the brain and the way that heart rate is regulated by the brain. The study also seeks to understand whether having depression changes the way that emotions and heart rate are regulated.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 years
* Able to understand and provide informed consent
* Male and female

Depressed Subjects:

* Current diagnosis of major depressive disorder (MDD) and currently in an major depressive episode (MDE)
* Quick Inventory of Depressive Symptomology (QIDS-SR16) score of 11 or greater
* Anticipated treatment with ketamine infusion for depression

Exclusion Criteria:

* Current daily use of tricyclic antidepressants
* Current diagnosis of cardiac arrhythmia or heart failure
* Pregnancy
* Current use of cardiac medications of the class beta-blockers
* Current treatment with deep brain stimulation for any reason

Healthy Controls:

* Current psychiatric treatment, including use of antidepressants or daily use of anxiolytic medication

Depressed Subjects:

* Previous history of ketamine infusion for depression
* Psychotic symptoms
* Active co-morbid psychiatric diagnosis including anxiety disorder or personality disorder that significantly affects the current clinical condition, as determined by medical records

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Change in heart rate variability (HRV, also called RSA) | Baseline, Post-Video Task Session 1 (30 minutes)
  HRV is measured as the variations of the time interval between two consecutive cardiac beats registered by means of electrocardiogram (EKG). Change is the difference from between HRV at baseline and after video task.
Change in heart rate variability (HRV, also called RSA) | Baseline, Post-Imaginal Task Session 1 (6 minutes)
  HRV is measured as the variations of the time interval between two consecutive cardiac beats registered by means of electrocardiogram (EKG). Change is the difference from between HRV at baseline and after the imaginal task.
Change in heart rate variability (HRV, also called RSA) | Baseline, Post-Video Task Session 2 (30 minutes)
  HRV is measured as the variations of the time interval between two consecutive cardiac beats registered by means of electrocardiogram (EKG). Change is the difference from between HRV at baseline and after video task one week post-infusion.
Change in heart rate variability (HRV, also called RSA) | Baseline, Post-Imaginal Task Session 2 (6 minutes)
  RSA is measured by changes in the R-R interval (time between two of the distinctive, large, upward "R" spikes on an electrocardiogram (EKG)) synchronized with respiration. Change is the difference from between RSA at baseline and after imaginal task one week post-infusion.

SECONDARY OUTCOMES:
Mean values of positive emotional expressions | Post-Video Task Session 1 (30 minutes)
  Automated analysis of video data of facial expressions will be carried out using iMotions software (iMotions Inc, Cambridge, MA). This software can calculate the probability of expression of certain emotional states (e.g. neutral, positive, negative).
Mean values of positive emotional expressions | Post-Imaginal Task Session 1 (6 minutes)
  Automated analysis of video data of facial expressions will be carried out using iMotions software (iMotions Inc, Cambridge, MA). This software can calculate the probability of expression of certain emotional states (e.g. neutral, positive, negative).
Mean values of negative emotional expressions | Post-Video Task Session 1 (30 minutes)
  Automated analysis of video data of facial expressions will be carried out using iMotions software (iMotions Inc, Cambridge, MA). This software can calculate the probability of expression of certain emotional states (e.g. neutral, positive, negative).
Mean values of negative emotional expressions | Post-Imaginal Task Session 1 (6 minutes)
  Automated analysis of video data of facial expressions will be carried out using iMotions software (iMotions Inc, Cambridge, MA). This software can calculate the probability of expression of certain emotional states (e.g. neutral, positive, negative).
Mean values of positive emotional expressions | Post-Video Task Session 2 (30 minutes)
  Automated analysis of video data of facial expressions will be carried out using iMotions software (iMotions Inc, Cambridge, MA). This software can calculate the probability of expression of certain emotional states (e.g. neutral, positive, negative).
Mean values of positive emotional expressions | Post-Imaginal Task Session 2 (6 minutes)
  Automated analysis of video data of facial expressions will be carried out using iMotions software (iMotions Inc, Cambridge, MA). This software can calculate the probability of expression of certain emotional states (e.g. neutral, positive, negative).
Mean values of negative emotional expressions | Post-Video Task Session 2 (30 minutes)
  Automated analysis of video data of facial expressions will be carried out using iMotions software (iMotions Inc, Cambridge, MA). This software can calculate the probability of expression of certain emotional states (e.g. neutral, positive, negative).
Mean values of negative emotional expressions | Post-Imaginal Task Session 2 (6 minutes)
  Automated analysis of video data of facial expressions will be carried out using iMotions software (iMotions Inc, Cambridge, MA). This software can calculate the probability of expression of certain emotional states (e.g. neutral, positive, negative).
Mean activation of muscle action units | Post-Video Task Session 1 (30 minutes)
  Automated analysis of video data of facial expressions will be carried out using iMotions software (iMotions Inc, Cambridge, MA). This software can calculate the activation of facial muscle action units.
Mean activation of muscle action units | Post-Imaginal Task Session 1 (6 minutes)
  Automated analysis of video data of facial expressions will be carried out using iMotions software (iMotions Inc, Cambridge, MA). This software can calculate the activation of facial muscle action units associated with smiling.
Mean activation of muscle action units | Post-Video Task Session 2 (30 minutes)
  Automated analysis of video data of facial expressions will be carried out using iMotions software (iMotions Inc, Cambridge, MA). This software can calculate the activation of facial muscle action units associated with smiling.
Mean activation of muscle action units | Post-Imaginal Task Session 2 (6 minutes)
  Automated analysis of video data of facial expressions will be carried out using iMotions software (iMotions Inc, Cambridge, MA). This software can calculate the activation of facial muscle action units associated with smiling.
Change in heart rate | Baseline, Post-Video Task Session 1 (30 minutes)
  Heart rate will be measured with the electrocardiogram (EKG) and recorded in beats per minute. Change is the difference from between heart rate at baseline and after the video task.
Change in heart rate | Baseline, Post-Imaginal Task Session 1 (6 minutes)
  Heart rate will be measured with the electrocardiogram (EKG) and recorded in beats per minute. Change is the difference from between heart rate at baseline and after the imaginal task.
Change in heart rate | Baseline, Post-Video Task Session 2 (30 minutes)
  Heart rate will be measured with the electrocardiogram (EKG) and recorded in beats per minute. Change is the difference from between heart rate at baseline and after the video task one week post-infusion.
Change in heart rate | Baseline, Post-Imaginal Task Session 2 (6 minutes)
  Heart rate will be measured with the electrocardiogram (EKG) and recorded in beats per minute. Change is the difference from between heart rate at baseline and after the imaginal task one week post-infusion.
Change in skin conductance response (SCR) | Baseline, Post-Video Task Session 1 (30 minutes)
  The skin conductance will be measured between two leads attached to the participant's the left and right palms which records electrodermal measures. Change is the difference from between SCR at baseline and after the video task.
Change in skin conductance response (SCR) | Baseline, Post-Imaginal Task Session 1 (6 minutes)
  The skin conductance will be measured between two leads attached to the participant's the left and right palms which records electrodermal measures. Change is the difference from between SCR at baseline and after the imaginal task.
Change in skin conductance response (SCR) | Baseline, Post-Video Task Session 2 (30 minutes)
  The skin conductance will be measured between two leads attached to the participant's the left and right palms which records electrodermal measures. Change is the difference from between SCR at baseline and after the video task one week post-infusion.
Change in skin conductance response (SCR) | Baseline, Post-Imaginal Task Session 2 (6 minutes)
  The skin conductance will be measured between two leads attached to the participant's the left and right palms which records electrodermal measures. Change is the difference from between SCR at baseline and after the imaginal task one week post-infusion.
Change in respiration rate | Baseline, Post-Video Task Session 1 (30 minutes)
  The respiration rate will be measured by the respiration monitor belt and recorded as number of breaths per minute. Change is the difference from between respiration rate at baseline and after the video task.
Change in respiration rate | Baseline, Post-Imaginal Task Session 1 (6 minutes)
  The respiration rate will be measured by the respiration monitor belt and recorded as number of breaths per minute. Change is the difference from between respiration rate at baseline and after the imaginal task.
Change in respiration rate | Baseline, Post-Video Task Session 2 (30 minutes)
  The respiration rate will be measured by the respiration monitor belt and recorded as number of breaths per minute. Change is the difference from between respiration rate at baseline and after the video task one week post-infusion.
Change in respiration rate | Baseline, Post-Imaginal Task Session 2 (6 minutes)
  The respiration rate will be measured by the respiration monitor belt and recorded as number of breaths per minute. Change is the difference from between respiration rate at baseline and after the imaginal task one week post-infusion.
Change in pulse rate | Baseline, Post-Video Task Session 1 (30 minutes)
  The peripheral pulse rate will be measured by pulse oximeters placed on one finger on the left and right hands. Change is the difference from between pulse rate at baseline and after the video task.
Change in pulse rate | Baseline, Post-Imaginal Task Session 1 (6 minutes)
  The peripheral pulse rate will be measured by pulse oximeters placed on one finger on the left and right hands. Change is the difference from between pulse rate at baseline and after the imaginal task.
Change in pulse rate | Baseline, Post-Video Task Session 2 (30 minutes)
  The peripheral pulse rate will be measured by pulse oximeters placed on one finger on the left and right hands. Change is the difference from between pulse rate at baseline and after the video task one week post-infusion.
Change in pulse rate | Baseline, Post-Imaginal Task Session 2 (6 minutes)
  The peripheral pulse rate will be measured by pulse oximeters placed on one finger on the left and right hands. Change is the difference from between pulse rate at baseline and after the imaginal task one week post-infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Crowell, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - 12 Executive Park Drive, Atlanta, Georgia
  - Emory University at Wesley Woods Hospital, Atlanta, Georgia